CLINICAL TRIAL: NCT06548776
Title: Establishing Daily Applicable Parameters for Using Magnetic Resonance Spectroscopy of Spinal Cord
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2024-0249; NCI-2024-06761 (Other: NCI-CTRP Clinical Trials Registry)
Record Dates: First submitted 2024-08-08; First posted 2024-08-12 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Spinal Cord
MeSH Terms: interventions — Positron-Emission Tomography; Radionuclide Imaging

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Healthy Volunteers (Experimental): Participants will be recruited from DI volunteer pool to implement MRS spine on.
  Interventions: Diagnostic Test: Magnetic Resonance Spectroscopy (MRS) Scan
- Patients (Experimental): Participants will be recruited from DI volunteer pool to implement MRS spine on.
  Interventions: Diagnostic Test: Magnetic Resonance Spectroscopy (MRS) Scan

INTERVENTIONS:
Diagnostic Test: Magnetic Resonance Spectroscopy (MRS) Scan — Participants will receive MRS Scan

SUMMARY:
To learn if MRS can effectively assess spinal cord lesions.

DETAILED DESCRIPTION:
Primary Objective:

Establish the feasibility and spectrum of MRS for adult patients while mapping the total spine spectrum at short TEs to allow for future comparison with patients to assess spinal cord lesions malignant potential and grade.

Secondary Objective:

Test success of the spectrum by implementing the protocol on 3 low volume LMD receiving LMD receiving CSI. This will allow us to test reproducibility of the protocol and test effect of radiation on spinal cord at different time frames. This will serve as secondary data for subsequent trials targeting functional statues after radiation and tumor grading predictability of MRS.

ELIGIBILITY:
Inclusion Criteria:

Volunteers:

* Adults > 18 years
* Healthy with no malignancy, demyelinating disease, back pain, degenerative disease, or spinal cord lesions.
* Consent able patients.

Patients with low volume LMD to receive treatment CNS radiation:

* Adults > 18 years old.
* MR or CSF with evidence of LMD.
* Patients to receive CSI as part of standard treatment of LMD disease.
* Consent able patients, willingness and ability to comply with the study procedures.
* No spinal cord lesions only LMD disease
* Recruitment by radiation oncology faculty in consultation with Dr. De. . .

Exclusion Criteria:

Volunteers:

* Age < 18 years
* Pregnant or breastfeeding individuals.
* History of cancer.
* History of spinal cord lesions including malignant, demyelinating, or inflammatory.
* History of prior spinal surgery.
* History of implantable devices.
* History of MR claustrophobia.
* Degenerative disease or spinal/back pain including myelopathy and radiculopathy.
* Scoliosis.

Patients with LMD:

* Age < 18 years
* History of spinal cord lesions including malignant, demyelinating, or inflammatory.
* History of prior spinal surgery.
* History of implantable devices.
* History of MR claustrophobia.
* Degenerative disease or spinal/back pain including myelopathy and radiculopathy.
* Scoliosis.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 13 (Estimated)
Dates: Start 2024-09-04 (Actual); Primary Completion 2026-07-31 (Estimated); Study Completion 2028-07-31 (Estimated)

PRIMARY OUTCOMES:
Safety and Adverse Events (AEs) | Through study completion; an average of 1 year.
  Incidence of Adverse Events, Graded According to National Cancer Institute Common Terminology Criteria for Adverse Events (NCI CTCAE)

CONTACTS AND LOCATIONS:
Overall Officials: Rami Eldaya, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center Website — http://www.mdanderson.org